CLINICAL TRIAL: NCT01447732
Title: Two-Part, Open-Label, Multi-Center Phase 1 Study of Monoclonal Antibody CEP-37250/KHK2804 in Subjects With Advanced Solid Tumors
Brief Title: Phase 1 Study of CEP-37250/KHK2804 in Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Collaborators: Teva Pharma (Industry); Kyowa Hakko Kirin Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEP-37250/KHK2804-001
Record Dates: First submitted 2011-09-30; First posted 2011-10-06 (Estimated); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Solid Tumour; Adenocarcinoma of the Colorectal; Adenocarcinoma of the Pancreas
Keywords: Monoclonal antibody (Mab); Antibody dependent cellular cytotoxicity (ADCC); Complement-dependent toxicity (CDC); Non-fucosylated immunoglobulin G
MeSH Terms: conditions — Mycobacterium Infections, Nontuberculous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1 (Experimental): Dose escalation in subjects with advanced solid tumors with Part 1 which includes intervention of CEP-37250/KHK2804
  Interventions: Drug: CEP-37250/KHK2804
- Part 2 (Experimental): Subjects with colorectal or pancreatic cancer Part 2 which includes intervention of CEP-37250/KHK2804
  Interventions: Drug: CEP-37250/KHK2804

INTERVENTIONS:
Drug: CEP-37250/KHK2804 — Part 1 is based on the CEP-37250/KHK2804 tolerability and safety data from three subjects enrolled in a cohort, enrollment at the next dose level or additional subjects into the ongoing cohort will occur based upon the number subjects with DLT at a given dose level. Dose depends on subject's body weight. Part 1 includes intervention of CEP-37250/KHK2804.
  Part 2 will receive CEP-37250/KHK2804 at a dose to be determined following completion of Part 1.
  Other Names: KHK2804

SUMMARY:
This is a two-part, Phase 1 open label, multi-center, dose escalation study of CEP-37250/KHK2804 as monotherapy in subjects with advanced solid tumors who no longer respond to standard therapy or for whom no standard therapy is available.

DETAILED DESCRIPTION:
The study will be conducted in two parts. In Part 1, a standard 3+3 designed dose escalation phase, subjects will receive CEP-37250/KHK2804, administered iv, once every week. A treatment cycle will consists of total of four doses per cycle. Part 2 of the study will enroll subjects with either colon cancer or pancreatic cancer to receive CEP-37250/KHK2804 at a dose to be determined following completion of Part 1.

All subjects will receive study therapy until disease progression, the development of unacceptable toxicity, noncompliance or withdrawal of consent by the subject, or Investigator decision, up to a maximum of six cycles (approximately six months). After six cycles of CEP-37250/KHK2804 therapy, the subject may continue to receive CEP-37250/KHK2804 after discussion with the Sponsor and determination that the subject is experiencing a best response of at least stable disease (SD) and is not experiencing any unacceptable toxicities or dose limiting toxicities (DLTs).

ELIGIBILITY:
Inclusion Criteria:

* Adequate hepatic, renal, and hematologic function;
* Life expectancy > 3 months;
* Part 1 and 2: The subject has histopathologically or cytologically documented, measurable, unresectable, locally advanced primary or recurrent, metastatic solid tumor, locally advanced primary or recurrent, metastatic pancreatic adenocarcinoma and must have received at least one prior treatment regimen containing gemcitabine or 5-FU, and locally advanced primary or recurrent, metastatic colon adenocarcinoma.

Exclusion Criteria:

* Parts 1 and 2:

  1. Malignant melanoma, Merkel cell cancer, small cell lung cancer, lymphoepithelial carcinoma, malignant mesothelioma, GIST, Hodgkin and NHL, thymoma, neuroendocrine, neuronal tumors, and sarcomas. This list of excluded tumors may be modified as additional research findings become available on target antigen expression;
  2. The subject has received anti-cancer chemotherapy, hormonal therapy, radiotherapy, immunotherapy, or investigational agents within 4 weeks (6 weeks for mitomycin C and nitrosoureas) prior to the first dose of CEP-37250/KHK2804;
  3. The subject has received monoclonal antibodies of any type or for any form of disease within 4 weeks of the first dose of CEP-37250/KHK2804;
  4. Major surgery within 4 weeks prior to the first dose;
  5. Known symptomatic brain metastases (screening magnetic resonance imaging (MRI) of the brain is only required when there is clinical suspicion of central nervous system [CNS] involvement or past history of treated brain metastasis). Subjects with treated brain metastasis (radiotherapy and/or surgery) will be eligible if they:
* Have completed treatment for their brain metastasis > 4 weeks prior to scheduled study treatment start date;
* Are neurologically stable;
* Are on corticosteroids in doses no greater than physiological replacement (e.g., dexamethasone < 1.5 mg/day); and
* Have a screening MRI scan of the brain that specifically verifies no evidence of CNS hemorrhage and no active gadolinium enhancing lesions;
* Subjects with primary brain/CNS malignancy (e.g., gliomas, lymphomas) are excluded.

  * Hypersensitivity reaction to monoclonal antibodies, other therapeutic proteins, or allergy to any component of the CEP-37250/KHK2804 finished drug and the reaction could not be controlled or prevented on subsequent infusion with standard therapies such as antihistamines, 5-HT3 antagonists, or corticosteroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2011-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Adverse Event collection and assessment will be done for all 74 potentially treated subjects. | at least 30 days or up to 12 weeks
  The safety of CEP-37250/KHK2804 will be determined by reported adverse events (AEs), changes in the physical examinations, vital laboratory evaluations, and treatment discontinuations due to toxicity.

SECONDARY OUTCOMES:
To assess PK parameters which include: area under the plasma concentration versus time curve (AUC), peak plasma concentration (Cmax), t 1/2 and CL of CEP-37250/KHK2804. | at least 30 days or up to 12 weeks
  Participating subjects will have serial blood samples taken to determine the PK profile of study drug.
To screen for the development of antibodies against CEP-37250/KHK2804 (immunogenicity) | at least 30 days or up to 12 weeks
  Subjects will have serial blood samples to check for the developments of anti-CEP-37250/KHK2804 antibodies.
To evaluate preliminary efficacy (overall response (Objective response rate(ORR; Complete Response(CR)+Partial Response(PR) and clinical benefit rate(CR+PR+stable disease(SD)). | up to 30 days or up to 12 weeks
  Tumor measurements and disease response assessments will be performed on all participating subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Tirgan, MD, Study Director — Kyowa Hakko Kirin Pharma, Inc.

REFERENCES:
- [Derived] Mita MM, Nemunaitis J, Grilley-Olson J, El-Rayes B, Bekaii-Saab T, Harvey RD, Marshall J, Zhang X, Strout V. Phase 1 Study of CEP-37250/KHK2804, a Tumor-specific Anti-glycoconjugate Monoclonal Antibody, in Patients with Advanced Solid Tumors. Target Oncol. 2016 Dec;11(6):807-814. doi: 10.1007/s11523-016-0449-2. PMID 27457707